CLINICAL TRIAL: NCT05503849
Title: Born In Guangzhou Intervention Study
Acronym: BIGIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Department of Women's Health, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022390B00
Record Dates: First submitted 2022-08-09; First posted 2022-08-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Outcomes; Child Development; Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive management during pregnancy (Experimental): A combination of dietary, physical activity and lifestyle modification.
  Interventions: Behavioral: Lifestyle modification
- Standard Care (No Intervention): No additional intervention beyond standard care procedure.

INTERVENTIONS:
Behavioral: Lifestyle modification — This lifestyle modification aiming to provide proactive health management during pregnancy, which contains the following: 1) balanced dietary intake based on the Chinese Dietary Guideline; 2) sufficient physical activity; 3) changes in lifestyles (e.g. sleep, sun exposure etc.)
  Arms: Proactive management during pregnancy

SUMMARY:
The main objective of this study is to test the efficacy of an intervention package (dietary, physical and lifestyle modification) during pregnancy in improving the clinical outcomes of mother-infant dyads.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending prenatal care at Guangzhou Women and Children's Medical Center (GWCMC) <20 weeks' gestation
* Pregnant women plan to deliver at GWCMC
* Pregnant women intend to reside in Guangzhou for at least 3 years

Exclusion Criteria:

* Multiple pregnancies
* Existing medical conditions (uncontrolled diabetes, hypertension or thyroid disease; other serious cardiovascular diseases, respiratory or systematic disorders)
* Use of drugs (aspirin, metformin, low molecular weight heparin)
* Women with reading and/or writing difficulties
* Women with serious mental disorders
* Women with eating disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1160 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Maternal gestational weight change | From pregnancy until one month postpartum
  Maternal weight prior to pregnancy (or within 8 weeks of pregnancy), at around 20, 26, 32 weeks' gestation, before delivery and one month postpartum will be determined by digital scales, changes in maternal weight during pregnancy will be recorded in kg.
Newborn size | Day 1 after birth
  Weight (kg) will be measured with digital scales and height/length (cm) will be measured in supine with tape, comparing against reference to derived gestational age and sex-specific growth parameter Z-scores. To identify whether the neonates was small/appropriate/large for gestational age.
Neonatal skinfold thickness (at birth) | Day 1 after birth
  Measured with skinfold caliper, a summation of skinfold thickness at several body sites including triceps, biceps, subscapular, suprailiac and thigh, will be derived in cm.
Maternal blood lipid profile postpartum (3 years) | Three years after delivery
  Measured by autoanalyzer, total lipids (total cholesterol, triglycerides, high/low density protein cholesterol) expressed in mmol/L.
Maternal blood glucose profile postpartum (3 years) | Three years after delivery
  Measured by autoanalyzer, blood glucose level in mmol/L.
Maternal blood insulin profile postpartum (3 years) | Three years after delivery
  Measured by commercial ELIZA kit, total and free insulin in pmol/L.
Child blood lipid profile (3 years) | At three years of age
  Measured by autoanalyzer, total lipids (total cholesterol, triglycerides, high/low density protein cholesterol) expressed in mmol/L.
Child blood glucose profile (3 years) | At three years of age
  Measured by autoanalyzer, blood glucose level in mmol/L.
Child blood insulin profile (3 years) | At three years of age
  Measured by commercial ELIZA kit, total and free insulin in pmol/L.
Child growth parameters (3 years) | At three years of age
  Weight measured with digital scales in kg, length measured in standing position in cm, using weight and length to derived body mass index, comparing against age and sex-specific references for Z-score.
Incidence of pregnancy complications | From 20 weeks' gestation until one month postpartum
  Incidence of physician-diagnosed pregnancy complications, including gestational diabetes mellitus, hypertensive disorders

SECONDARY OUTCOMES:
Child skinfold thickness (6 months) | At six months of age
  Measured with skinfold caliper, a summation of skinfold thickness at several body sites including triceps, biceps, subscapular, suprailiac and thigh, will be derived in cm.
Child skinfold thickness (1 year) | At one year of age
  Measured with skinfold caliper, a summation of skinfold thickness at several body sites including triceps, biceps, subscapular, suprailiac and thigh, will be derived in cm.
Child skinfold thickness (3 years) | At three years of age
  Measured with skinfold caliper, a summation of skinfold thickness at several body sites including triceps, biceps, subscapular, suprailiac and thigh, will be derived in cm.
Child skinfold thickness (6 years) | At six years of age
  Measured with skinfold caliper, a summation of skinfold thickness at several body sites including triceps, biceps, subscapular, suprailiac and thigh, will be derived in cm.
Child growth parameters (6 months) | At six months of age
  Weight measured with digital scales in kg, length measured with tape in supine position in cm, using weight and length to derived body mass index, comparing against age and sex-specific references for Z-score.
Child growth parameters (1 year) | At one year of age
  Weight measured with digital scales in kg, length measured with tape in supine position in cm, using weight and length to derived body mass index, comparing against age and sex-specific references for Z-score.
Child growth parameters (6 years) | At six years of age
  Weight measured with digital scales in kg, length measured in standing position in cm, using weight and length to derived body mass index, comparing against age and sex-specific references for Z-score.
Child blood lipid profile (6 years) | At six years of age
  Measured by autoanalyzer, total lipids (total cholesterol, triglycerides, high/low density protein cholesterol) expressed in mmol/L
Child blood sugar profile (6 years) | At six years of age
  Measured by autoanalyzer, blood glucose level in mmol/L.
Child blood insulin profile (6 years) | At six years of age
  Measured by commercial ELIZA kit, total and free insulin in pmol/L.
Neurological development of child (1 year) | At one year of age
  Assessed by using Gesell testing, which measures the child's cognitive, language, motor (gross & fine) and social-emotional responses. Higher score in each domain is desired, there is no upper limit. Overall score of less than 86 indicates suspected developmental retardation.
Neurological development of child (3 years) | At three years of age
  Assessed by Ages & Stages Questionnaires, including adaptive, motor (gross & fine), language, and social function domains, overall score being less than -2SD of age specific mean indicates suspected developmental retardation.
Maternal hand grip strength during pregnancy | Between 32-34 weeks' gestation
  Measured by high precision digital hand dynamometer, in kg
Maternal hand grip strength after delivery | At one month postpartum
  Measured by high precision digital hand dynamometer, in kg
Maternal body composition postpartum | At one month postpartum
  Measured by dual-energy X-ray absorptiometry by trained physician, fat mass (kg), fat free mass (kg), and relative proportion (%) and distribution of fat mass will be described.
Maternal blood lipid profile postpartum (6 years) | Six years after delivery
  Measured by autoanalyzer, total lipids (total cholesterol, triglycerides, high/low density protein cholesterol) expressed in mmol/L.
Maternal blood sugar profile postpartum (6 years) | Six years after delivery
  Measured by autoanalyzer, blood glucose level in mmol/L.
Maternal blood insulin profile postpartum (6 years) | Six years after delivery
  Measured by commercial ELIZA kit, total and free insulin in pmol/L.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fuying Campus, Guangzhou Women and Children's Medical Center, Guangzhou Medical University, Guangzhou, China, Guangzhou
  - Zhujiang new town campus, Guangzhou Women and Children's Medical Center, China, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694